CLINICAL TRIAL: NCT01900886
Title: Prospective Observational Study to Assess Personality Disorders in Prison Populations for Hepatitis C Treatment. "
Brief Title: Epidemiological Study to Evaluate Personality Disorders in Prison Populations in Treatment for Hepatitis C
Acronym: Perseo
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Grupo de Enfermedades Infecciosas de la Sociedad Española de Sanidad Penitenciaria (Other)
Responsible Party: Sponsor
Other Study IDs: GEI-HCC-2010-01
Record Dates: First submitted 2013-07-08; First posted 2013-07-17 (Estimated); Last update posted 2013-07-17 (Estimated); Status verified 2010-12

CONDITIONS: Hepatitis C, Chronic; Personality Disorders in Prison
Keywords: prison, disorder, hepatitis c
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pegasys, injection subcutaneous: Hepatitis C Virus (HCV) patients monoinfected or coinfected, all genotypes, treatment naive to Peginterferon alfa-2a and Ribavirin (RBV)
  Interventions: Other: Peginterferon alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Other: Peginterferon alfa-2a — Treatment as usual clinical practice
  Other Names: Pegasys
Drug: Ribavirin — Treatment as usual clinical practice
  Other Names: Copegus

SUMMARY:
Primary objective: Evaluate the prevalence of personality disorders in patients starting treatment for hepatitis C in the prison and determine their influence on the evolution of the disease.

DETAILED DESCRIPTION:
Secondary objectives:

* Describe the management of patients with personality disorders on treatment for hepatitis C in the prison.
* Describe the characteristics of patients who discontinue the treatment and the reasons for stratifying by the presence of personality disorders.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age.
* Patients with expected prison stay beyond the duration of follow-up period of the study.
* Patients with chronic HCV infection and detectable viral load to initiate treatment with standard therapy.
* Patients their written informed consent to participate in the study.

Exclusion Criteria:

* Patients previously treated with Interferon (IFN) and Ribavirin (RBV).
* Patients can not read or understand a written questionnaire at the discretion of the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients with chronic hepatitis C mono-or co-infected with HIV.
Sampling Method: Non-Probability Sample
Enrollment: 263 (Estimated)
Dates: Start 2010-12; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Sustained Viral Response (SVR) | RNA-VHC at weeks 24 or 48

CONTACTS AND LOCATIONS:
Overall Officials: Andres Marco, Medicine, Principal Investigator — Centro Penitenciario de Hombres de Barcelona. Prisión Modelo
Locations (11):
- Spain (11):
  - Centro Penitenciario de El Acebuche, Almería, Almeria
  - Centro Penitenciario de Badajoz, Badajoz, Badajoz
  - Centro Penitenciario El Puerto III, Jerez de la Frontera, Cadiz
  - Centro Penitenciario Las Palmas, Las Palmas de Gran Canaria, Canary Islands
  - Centro Penitenciario de Tenerife, Santa Cruz de Tenerife, Canary Islands
  - Centro Penitenciario de Cordoba, Córdoba, Cordoba
  - Centro Penitenciario de Albolote, Albolote, Granada
  - Centro Penitenciario Jaen, Jaén, Jaen
  - Centro Penitenciario de Topas, Salamanca, Salamanca
  - Centro Penitenciario Sevilla I, Seville, Sevilla
  - Centro Penitenciario Ocaña I, Ocaña, Toledo

REFERENCES:
- [Derived] Marco A, Anton JJ, Trujols J, Saiz de la Hoya P, de Juan J, Faraco I, Cayla JA; Perseo Group. Personality disorders do not affect treatment outcomes for chronic HCV infection in Spanish prisoners: the Perseo study. BMC Infect Dis. 2015 Aug 19;15:355. doi: 10.1186/s12879-015-1102-x. PMID 26286450